CLINICAL TRIAL: NCT04471532
Title: Promotion and Support for Physical Activity Maintenance Post Total Hip Arthroplasty (PANORAMA). A Pragmatic, Randomized, Controlled, Trial.
Brief Title: Promotion and Support for Physical Activity Maintenance Post Total Hip Arthroplasty
Acronym: PANORAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); Helsefonden, Denmark (Unknown); Hartmann Fonden (Other)
Responsible Party: Principal Investigator, Theresa Bieler, Research Therapist, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19050820
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Exercise; Motivation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, randomized, controlled, assessor- and statistician- blinded trial with two parallel groups; an intervention group receiving a behavior change intervention and a control group receiving no intervention.
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be blinded to group allocation and previous results and the participants are requested not to disclose their allocation when outcomes are assessed 6 and 12 months after surgery.
  The biostatistician who perform the data analyses and validate the results will also be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior change intervention (Experimental): A 3-month behavior change intervention i.e. one initial, face-to-face, physical activity counselling and two telephone-assisted counselling.
  Interventions: Behavioral: Behavior change intervention
- Control (No Intervention): No attention

INTERVENTIONS:
Behavioral: Behavior change intervention — It is a 3-month, multimodal, minimal contact, pedometer-driven, behavior change intervention to promote and support physical activity, that is initiated 3 months after THA. There is one initial, physiotherapist-led, face-to-face, physical activity counselling including 1) a brief motivational interviewing regarding physical activity, 2) patient education regarding physical activity after THA including recommendations and safety based on an "orthopedic surgeon guided" video and leaflet, 3) handling out pedometer and educational material i.e. a practice-oriented leaflet with advice on how to use a pedometer, a step-calendar and goal setting as well as strategies to incorporate physical activity into daily life. This initial counselling is followed by two, physiotherapist-led, telephone-assisted counselling after respectively three and seven weeks.
  Arms: Behavior change intervention

SUMMARY:
Total hip arthroplasty (THA) is considered an efficacious procedure for relieving pain and disability in patients with hip osteoarthritis. However, 6-12 months post-surgery physical activity level is unchanged compared to pre-surgery and still considerably lower than that of healthy peers. Increasing physical activity after THA may enhance the outcome of the THA because a graded relationship between physical activity level and functional performance has been documented. Six-8 months after THA physical function is only recovered to about 80% of that of healthy peers and older adults still seem to be at increased risk of frailty. Furthermore, these patients continue to impose higher healthcare costs than an age- and sex-matched reference population which potentially could be related to the functional status that is not completely regained. Finally, patients with hip osteoarthritis can have extensive comorbidity thus increasing physical activity after THA could be a simple and relatively inexpensive method for improving general health, which in turn may decrease healthcare costs.

The reasons for the lack of increase in physical activity despite increased capability after THA are unknown but it may be related to the sedentary behavior adopted by the patients prior to surgery and uncertainty. A systematic review has illuminated that patient-reported barriers to engaging in physical activity after THA are largely related to limited or inadequate information or education culminating in uncertainty about 'doing the right thing' for both the individual's recovery and the longevity of the joint replacement.

Few studies have investigated the effects of specific interventions to increase physical activity after THA. Promising results have been shown from physical activity sensors in combination with e.g. goal setting. None of these studies have addressed the patient-reported barriers to physical activity regarding uncertainty and limited education.

This trial aims to investigate the effect of adding a pedometer-driven, behavior change intervention to usual rehabilitation care 3 months after THA to increase physical activity compared to usual rehabilitation care alone (control). Outcomes are taken 3 (baseline), 6 (after the intervention period) and 12 months after THA (follow-up).

Hypothesis: the behavior change intervention will increase the proportion that completes ≥8,000 steps per day 6-month post-surgery to 50% versus 30% in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Home dwelling, independent and self-reliant adults
* Patients who has received primary total hip arthroplasty because of hip osteoarthritis
* Informed consent to participate

Exclusion Criteria:

* Planned joint arthroplasty in the lower extremities within the next 6 months
* Patients who are unable to read, understand and speak Danish
* Complications in relation to total hip arthroplasty e.g. dislocation, fracture or infection
* Any other condition that in the opinion of the investigator makes a potential participant unfit for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
The number of participants that complete ≥ 8,000 steps per day | 6 months after THA
  The mean number of steps completed per day assessed by an accelerometer during a 7-day period.

SECONDARY OUTCOMES:
The number of participants that complete ≥ 10,000 steps per day | 6 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.
Change from baseline in the 6-minute walk test | 6 months after THA
  The 6-minute walk test is a performance-based test of physical function which covers the domain ability to walk over longer distances. It is also a proxy measure of endurance/aerobic capacity. This test measures the walking distance completed in 6 minutes on a 30-m flat course. The participant is instructed to walk as far as possible in 6 minutes. The 6-minute walk test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in the 30-s chair-stand test | 6 months after THA
  The 30-s chair-stand test is a performance-based test of physical function which covers the domains: sitting and getting in/out of a seated position. It is also a proxy measure for assessing lower body muscle strength and power. This test measures number of chair stands completed in 30 seconds. The participant is instructed to complete as many chair stands as possible in 30 seconds with arms across the chest. The 30-s chair-stand test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in the stair-climb test | 6 months after THA
  The stair-climb test is a performance-based test of physical function which covers the domains: mobility and climbing. It is also a proxy measure for assessing lower extremity muscle strength and power and balance. This test measures the time (best of two trials) to ascend and descend a flight of 10 steps. The participant is instructed to ascend and descend the flight of stairs as fast as possible. The stair-climb test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in self-reported physical function | 6 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the function in daily living (ADL) subscale. The last week is taken into consideration when answering the 17 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in hip pain | 6 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the pain subscale. The last week is taken into consideration when answering the 10 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in the patients' assessment of global perceived effect | 6 months after THA
  The participants will be asked to compare their current global wellbeing with the pre-surgery state on a 200 mm visual analog scale with anchors being: -100 = "Much worse"; 0 = "No changes"; 100 = "Much better".
The mean number of steps per day | 6 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.
The number of participants that complete ≥ 5,000 steps per day | 6 and 12 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.
Health-related quality of life | 6 and 12 months after THA
  Assessed by the EuroQol 5-Dimension Questionnaire (EQ-5D-3L), a generic instrument with 5 questions that comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 3 levels: no problems, some problems, and extreme problems, where each dimension is assigned a score from 1 to 3, which can be converted into a single summary index value (based on the Danish EQ-5D Time Trade-Off (TTO) value set; 1 corresponds to the best possible health status, <0 represents the worst possible health status)

OTHER OUTCOMES:
The number of participants that complete ≥ 8,000 steps per day | 12 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.
The number of participants that complete ≥ 10,000 steps per day | 12 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.
Change from baseline in the 6-minute walk test | 12 months after THA
  The 6-minute walk test is a performance-based test of physical function which covers the domain ability to walk over longer distances. It is also a proxy measure of endurance/aerobic capacity. This test measures the walking distance completed in 6 minutes on a 30-m flat course. The participant is instructed to walk as far as possible in 6 minutes. The 6-minute walk test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in the 30-s chair-stand test | 12 months after THA
  The 30-s chair-stand test is a performance-based test of physical function which covers the domains: sitting and getting in/out of a seated position. It is also a proxy measure for assessing lower body muscle strength and power. This test measures number of chair stands completed in 30 seconds. The participant is instructed to complete as many chair stands as possible in 30 seconds with arms across the chest. The 30-s chair-stand test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in the stair-climb test | 12 months after THA
  The stair-climb test is a performance-based test of physical function which covers the domains: mobility and climbing. It is also a proxy measure for assessing lower extremity muscle strength and power and balance. This test measures the time (best of two trials) to ascend and descend a flight of 10 steps. The participant is instructed to ascend and descend the flight of stairs as fast as possible. The stair-climb test is included in a set of performance-based test recommended by the Osteoarthritis Research Society International that represents typical activities relevant to individuals following total joint arthroplasties.
Change from baseline in self-reported physical function | 12 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the function in daily living (ADL) subscale. The last week is taken into consideration when answering the 17 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in hip pain | 12 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the pain subscale. The last week is taken into consideration when answering the 10 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in the patients' assessment of global perceived effect | 12 months after THA
  The participants will be asked to compare their current global wellbeing with the pre-surgery state on a 200 mm visual analog scale with anchors being: -100 = "Much worse"; 0 = "No changes"; 100 = "Much better".
Change from baseline in self-reported physical activity | 6 and 12 months after THA
  Assessed by the Physical Activity Scale for the Elderly (PASE) that assesses the level of physical activity (occupational, household and leisure activities) over a one-week period. The score range is 0-400 or more (lowest to highest physical activity-level).
Change from baseline in self-reported physical activity level | 6 and 12 months after THA
  Assessed by a question "How physically active are you now?" from the Copenhagen City Heart Study (level 1-4; 1 = almost entirely sedentary, 2 = light physical activity (PA) for 2-4 h per week, 3 = light PA >4 h per week or more vigorous PA for 2-4 h per week, 4 = more vigorous PA >4 h per week or regular heavy exercise or competitive sports several times per week).
Change from baseline in Health-related quality of life | 6 and 12 months after THA
  Assessed by the EuroQol 5-Dimension Questionnaire (EQ-5D-3L), a generic instrument with 5 questions that comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 3 levels: no problems, some problems and extreme problems and a separate 20cm visual analog scale with anchors being: 0="worst imaginable health state"; 100="best imaginable health state".
Change from baseline in self-efficacy for physical activity | 6 and 12 months after THA
  Assessed by the exercise self-efficacy scale, which consists of 5 questions concerning the confidence of perceived ability to participate in exercise despite barriers as bad mood, bad weather, tiredness or lack of time (total score range, 5-25, worst to best).
Change from baseline in task-specific self-efficacy | 6 and 12 months after THA
  Assessed in conjunction with the stair-climbing test. After a practice trial, the participants are asked to rate their level of certainty that they can complete the stair-climbing task 2, 4, 6, 8, and 10 times without stopping (total score 0-100 (worst to best)).
Change from baseline in outcome expectancy for physical activity | 6 and 12 months after THA
  Assessed by the Outcome expectancy for exercise scale (OEE-2), an interviewer administered questionnaire with 13 questions regarding both positive and negative expectations associated with exercise. A positive outcome expectancy subscale, a negative outcome expectancy subscale and a total score can be calculated (more positive outcome expectations for exercise with higher score).
Change from baseline in symptoms (other than pain) | 6 and 12 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the other symptoms subscale. The last week is taken into consideration when answering the 5 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in function in sport and recreation | 6 and 12 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the function in sport and recreation subscale. The last week is taken into consideration when answering the 4 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
Change from baseline in hip-related quality of life | 6 and 12 months after THA
  Assessed by the Hip disability and Osteoarthritis Outcome Score (HOOS), the hip-related quality of life subscale. The last week is taken into consideration when answering the 4 questions (5 Likert boxes) included in this subscale. A normalized score (0-100, worst to best) can be calculated.
The mean number of steps per day | 12 months after THA
  The mean number of steps completed per day assessed with an accelerometer during a 7-day period.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Bieler, PT, PhD, Study Director — Bispebjerg and Frederiksberg Hospital, Dept. of Physical & Occupational Therapy
Locations (1):
- Bispebjerg Hospital, Department of Physical & Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Proposal for data use should be addressed to theresa.bieler@regionh.dk. Data access in Denmark is under very strict juristic data protection law. Any possible access or sharing demands a part application to: The Danish Data Protection Agency and The Ethics Committee of the Capital Region. Only if the applications are approved data will be considered available for sharing. The authors will not be able to support this process and a prolonged process must be expected.
Supporting Information: SAP, Analytic Code
Time Frame: Statistical Analysis Plan (SAP) available from 19.12.23, Analytic Code unresolved
Access Criteria: Please read plan description

REFERENCES:
- [Derived] Bieler T, Magnusson SP, Siersma V, Rinaldo M, Schmiegelow MT, Beck T, Krifa AM, Kjaer BH, Palm H, Midtgaard J. Effectiveness of promotion and support for physical activity maintenance post total hip arthroplasty-study protocol for a pragmatic, assessor-blinded, randomized controlled trial (the PANORAMA trial). Trials. 2022 Aug 13;23(1):647. doi: 10.1186/s13063-022-06610-4. PMID 35964101

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04471532/SAP_000.pdf